CLINICAL TRIAL: NCT03317418
Title: Can Pregnancy be Predicted According to ATR-FTIR Spectrophotometry of Incubation Medium of Embryos in IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0071-17
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ATR-FTIR Spectrophotometry — Spectrometry imaging

SUMMARY:
The aim of this study is to examine the variability of culture media composition based on the ATR-FTIR (Attenuated Total Reflectance-Fourier Transform Infrared Spectroscopy) technique on the day of embryo transfer/vitrification. In addition, the study will explore whether variations detected in the culture medium can be linked to embryo quality and the chances of achieving pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatments with at least 4 embryos

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women attending the fertility clinic at Hillel Yaffe Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Spectrometry in embryo culture media | One year
  Definition of spectrometry in embryo culture media
Embryo quality | One year
  The spectrometry results will be linked to embryo quality through the linkage between spectrometry results as indicated on Absorbance Graph and embryo quality judged by accepted criteria

SECONDARY OUTCOMES:
Cycle outcomes | One year
  Prediction of pregnancy rates as linked to the spectrometry results of the culture media

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom Paz, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No